CLINICAL TRIAL: NCT02273557
Title: Bioavailability of Dipyridamole of Asasantin p.o. (Extended Release 200 mg Dipyridamole/25 mg ASA) in Three Experimental Formulations (Given BID Over 3 Days Each) Relative to the Standard Formulation After a run-in Phase (Persantine ER BID for 2 Days Each: 25 mg, 50 mg, 100 mg; 150 mg [Persantine®]; 200 mg Persantine/25 mg ASA [Asasantin ER] in Healthy Male Subjects. Four-way, Change-over, Randomised, Open
Brief Title: Bioavailability of Dipyridamole of Asasantin p.o. in Three Experimental Formulations Relative to the Standard Formulation in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9.163
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (4):
- Asasantin ER (new formulation I - low) (Experimental)
  Interventions: Drug: Asasantin ER (new formulation I - low)
- Asasantin ER (new formulation III - medium) (Experimental)
  Interventions: Drug: Asasantin ER (new formulation III - medium)
- Asasantin ER (new formulation II - high) (Experimental)
  Interventions: Drug: Asasantin ER (new formulation II - high)
- Asasantin ER (present commercial formulation) (Active Comparator)
  Interventions: Drug: Asasantin ER (present commercial formulation)

INTERVENTIONS:
Drug: Asasantin ER (new formulation I - low)
  Arms: Asasantin ER (new formulation I - low)
Drug: Asasantin ER (new formulation III - medium)
  Arms: Asasantin ER (new formulation III - medium)
Drug: Asasantin ER (new formulation II - high)
  Arms: Asasantin ER (new formulation II - high)
Drug: Asasantin ER (present commercial formulation)
  Arms: Asasantin ER (present commercial formulation)

SUMMARY:
The objective of this study was to compare the pharmacokinetics of dipyridamole in three different Asasantin ER batches (test) containing different amounts of retarding lacquers to the existing commercial product at steady state with BID treatment

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >=50 years
* BMI >=18.5 and <=29.9 kg/m2
* Able to communicate well with the investigator and to comply with study requirements
* Laboratory values within a clinically defined reference range

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial, (< 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 3 months prior to administration (at least 10 times the relevant elimination half-life) or during trial)
* Having had prescription medication 2 weeks prior to study drug administration or over the counter medication 1 week prior to study drug administration (at least 10 times the relevant elimination half-life)
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation or loss > 400 mL (< 1 month prior to administration or during the trial)
* Excessive physical activities (< 5 days prior to administration or during the trial)
* Any ECG value outside of the reference range of clinical relevance including, but not limited to QTcB > 480 ms or QRS interval > 110 ms
* History of any familial bleeding disorder
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-01; Primary Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Urinary excretion of dipyridamole | day 2, day 3
  represented by the sum of percentage of amount excreted from time zer0 to 10 h (%Ae 0-10 h), %Ae 10-24h

SECONDARY OUTCOMES:
Cmax urine (Maximum measured concentration of the analyte) | 0 to 3 hours after drug intake
  Urine collected fraction from 0 -3 hours as surrogate for Cmax
Cmin urine (Minimum measured concentration of the analyte) | 8- 10 hours after drug intake
  Urine collected fraction from 8 - 10 hours as surrogate for Cmin
%PTF urine (Peak trough fluctuation) | Up to 10 hours after drug intake
  Estimated from the difference of percentage amount excreted from 1 - 3 hours (%Ae (1-3hours) and %Ae (8-10 hours) divided by the average excretion rate over the total dosing interval
Number of subjects with adverse events | up to 23 days